CLINICAL TRIAL: NCT06816745
Title: Comparison of Physiological Effects of Standard and Modified High-Flow Oxygen Therapy in Tracheostomized Patients
Brief Title: Comparison of Physiological Effects of Two Types of High-Flow Oxygen Therapy in Tracheostomized Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024-158-002
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Critical Care; Oxygen Therapy; Tracheostomy
Keywords: high-flow tracheal oxygen; tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified high flow tracheal oxygen (Experimental): Modified high-flow tracheal oxygen with flow rates of 40L/ min and 60L/min will be performed in tracheostomized patients.
  Interventions: Procedure: Modified high flow tracheal oxygen
- Standard high flow tracheal oxygen (Experimental): Standard high-flow tracheal oxygen with flow rates of 40 L/min and 60 L/min will be performed in tracheostomized patients.
  Interventions: Procedure: Standard high flow tracheal oxygen

INTERVENTIONS:
Procedure: Modified high flow tracheal oxygen — Modified high-flow tracheal oxygen with flow rates of 40L/min and 60L/min will be performed.
  Arms: Modified high flow tracheal oxygen
Procedure: Standard high flow tracheal oxygen — Standard high-flow tracheal oxygen with flow rates of 40 L/min and 60 L/min will be performed.
  Arms: Standard high flow tracheal oxygen

SUMMARY:
High-flow nasal oxygen therapy offers benefits like precise oxygen delivery, flow-related positive end-expiratory pressure generation and improved lung function. High-flow oxygen therapy can be applied via tracheostomy as high-flow tracheal oxygen. While high-flow tracheal oxygen has been used to facilitate weaning, it has diminished physiological effects due to bypassing upper airways. To enhance its effectiveness, researchers developed a modified high-flow tracheal oxygen tube with a smaller expiratory end diameter to increase airway resistance and pressure. This is a prospective randomized crossover study that aims to compare the physiological effects of standard and modified high-flow oxygen therapy in tracheostomized patients.

DETAILED DESCRIPTION:
High-flow nasal oxygen therapy has been shown to provide several physiological benefits, including precise control of the fraction of inspired oxygen, generation of flow-related positive end-expiratory pressure, increased end-expiratory lung volume, improved oxygenation, and enhanced carbon dioxide elimination. It has been widely utilized in managing acute hypoxemic respiratory failure and preventing hypoxemia after extubation.

High-flow oxygen therapy can be applied via tracheostomy as high-flow tracheal oxygen. Previous studies have reported successful cases of using high-flow tracheal oxygen to facilitate weaning from prolonged mechanical ventilation in patients with restrictive and obstructive pulmonary disorders. However, compared to high-flow nasal oxygen, high-flow tracheal oxygen exhibits significantly diminished physiological effects due to the bypassing of the narrow nasopharynx, glottis, and upper airway, as well as a more open circuit.

To address this limitation, the investigators have developed a modified high-flow tracheal oxygen tube with a reduced expiratory end tube diameter. This modification aims to create higher expiratory resistance and airway pressure, thus simulating the physiological effects of high-flow nasal cannula. This is a prospective randomized crossover physiological trial designed to compare the effects of standard and modified high-flow oxygen therapy in tracheostomized patients. Key physiological parameters will be assessed, including airway pressure, end-expiratory lung volume, vital signs, oxygenation, and respiratory workload.

ELIGIBILITY:
Inclusion Criteria:

Tracheostomy with stable spontaneous breathing.

Exclusion Criteria:

1. Age younger than 18 years old
2. Pregnancy
3. Hemodynamic instability (mean arterial pressure <60 mmHg, heart rate >140 or <60 bpm)
4. Respiratory and oxygenation instability (respiratory rate > 35bpm or oxygen saturation measured by pulse oximetry <90%)
5. Neuromuscular diseases or phrenic nerve injury
6. Recent trauma or surgery to the trachea, esophagus, neck, chest, or stomach
7. Pneumothorax or placement of a chest drainage
8. Contraindication to electrical impedance tomography (EIT) (implantable defibrillator)
9. Anticipating withdrawal of life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean expiratory airway pressure | From enrollment to the end of treatment at 4 hours
  Mean expiratory airway pressure will be measured during standard and modified high-flow tracheal oxygen.
Positive end-expiratory pressure | From enrollment to the end of treatment at 4 hours
  Positive end-expiratory pressure will be measured during standard and modified high-flow tracheal oxygen.
Change of end-expiatory lung volume | From enrollment to the end of treatment at 4 hours
  Change of end-expiatory lung volume will be measured during standard and modified high-flow tracheal oxygen.

SECONDARY OUTCOMES:
Respiratory rate | From enrollment to the end of treatment at 4 hours
  Respiratory rate will be measured during standard and modified high-flow tracheal oxygen.
Tidal volume | From enrollment to the end of treatment at 4 hours
  Tidal volume will be measured during standard and modified high-flow tracheal oxygen.
End-tidal carbon dioxide | From enrollment to the end of treatment at 4 hours
  End-tidal carbon dioxide will be measured during standard and modified high-flow tracheal oxygen.
Pulse oxygen saturation | From enrollment to the end of treatment at 4 hours
  Pulse oxygen saturation will be measured during standard and modified high-flow tracheal oxygen.
Esophageal pressure-time product | From enrollment to the end of treatment at 4 hours
  Esophageal pressure-time product will be measured during standard and modified high-flow tracheal oxygen.
Tidal swing of esophageal pressure | From enrollment to the end of treatment at 4 hours
  Tidal swing of esophageal pressure will be measured during standard and modified high-flow tracheal oxygen.
Respiratory muscle pressure | From enrollment to the end of treatment at 4 hours
  Respiratory muscle pressure will be measured during standard and modified high-flow tracheal oxygen.
Dynamic transpulmonary pressure | From enrollment to the end of treatment at 4 hours
  Dynamic transpulmonary pressure will be measured during standard and modified high-flow tracheal oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No